CLINICAL TRIAL: NCT01118455
Title: An Open Randomized Trial to Assess the Efficacy and Safety of Vagus Nerve Stimulation (VNS) Versus New Anti-Epileptic Drug (AED) Treatment in Children With Refractory Seizures
Brief Title: Trial to Assess Vagus Nerve Stimulation Therapy vs. Anti-Epileptic Drug (AED) Treatment in Children With Refractory Seizures
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Insufficient enrollment
Sponsor: Cyberonics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Epilepsy (E)-06
Record Dates: First submitted 2010-05-05; First posted 2010-05-06 (Estimated); Results first posted 2014-06-26 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-06

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — Vagus Nerve Stimulation; Therapeutics; Anticonvulsants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vagus Nerve Stimulation (VNS) Therapy (Experimental): Vagus Nerve Stimulation (VNS) Therapy is delivered by an implantable device similar to a pacemaker that sends mild stimulation to the left vagus nerve to help improve seizure control.
  Interventions: Device: Vagus Nerve Stimulation (VNS) Therapy
- Anti-Epileptic Drug (AED) (Experimental): This arm will supply a comparison between VNS and new AEDs which is necessary to determine an overall treatment regimen for the 30% to 40% of patients who fail to respond to 2 AEDs.
  Interventions: Drug: Anti-Epileptic Drug (AED)

INTERVENTIONS:
Device: Vagus Nerve Stimulation (VNS) Therapy — Vagus Nerve Stimulation (VNS) Therapy is delivered by an implantable device similar to a pacemaker that sends mild stimulation to the left vagus nerve to help improve seizure control.
  Arms: Vagus Nerve Stimulation (VNS) Therapy
Drug: Anti-Epileptic Drug (AED) — Subject has tried at least 2 appropriate AEDs tested to tolerance or to blood levels at upper end of the target range of which at least 2 had been tolerated at normal doses.
  Arms: Anti-Epileptic Drug (AED)

SUMMARY:
This is a randomized study designed to compare long-term treatment outcomes in pediatric patients with refractory seizures treated with VNS (Vagus Nerve Stimulation) Therapy versus anti-epileptic drugs (AEDs). Seizure reduction, quality of life measures, and side effect profiles will be evaluated. The results of this study will provide controlled comparative data to better guide physicians in determining the best overall treatment strategy for patients with seizures who have failed initial AED therapy.

DETAILED DESCRIPTION:
This was a randomized, parallel group, multi-center study. Screening Visit (visit 1) Subjects, parents, and the investigator signed and dated the informed consent after which subject eligibility was checked. Eligible subjects were entered in the baseline period.

Baseline Period (between visits 1 and 2) Eligible subjects entered an 8-week baseline period during which a seizure count was done. During this period, subjects and caregivers were contacted on a regular basis to ensure up to date information collection.

At the end of the baseline period, subjects who continued to be eligible were stratified based on previous therapy history (Early: previously treated with 2 to 5 AEDs versus Non-early: previously treated with >5 AEDs). Within each stratification, the investigator randomized each subject to receive one of the 2 treatments (VNS Therapy treatment or AED treatment) at the end of visit 2 using a randomization schedule provided by an independent third party (Synergos).

Implantation/AED Treatment Initiation (visit 3) For subjects randomized to the AED arm, a new AED treatment was initiated and gradually increased to an effective dose in accordance with the investigator's discretion and the manufacturer's suggested guidelines.

Subjects randomized to the VNS treatment arm were implanted with the VNS Therapy System and allowed adequate surgical recovery according to usual clinical practice before initiation of treatment. A delay of 2 weeks between the end of the baseline period and surgery was authorized to allow practical organization of the implantation. Extension of this period was approved in advance by the Study Director or his delegate.

Treatment Ramp-up (between visits 3 and 4) This ramp-up period for both AEDs and VNS may have taken up to 9 weeks, ending at visit 4. Additional visits were scheduled outside of the study protocol to adequately accommodate Treatment Ramp-up as needed. Initiation of treatments as well as the ramp-up schedule was documented in the Case Report Forms.

Study Treatment Period The Study Treatment Period was 12 months (52 weeks) following visit 3 and including Treatment Ramp-up. Because this study was designed to compare the natural course of treatment, changes in the study AED dose (for the AED group) or VNS stimulation parameters (for the VNS Therapy group) were allowed as clinically indicated during the Study Treatment Period. The protocol allowed approximately a 10% increase in baseline AED to allow for an increase in growth of the patient in the VNS arm.

Study End At the end of the study, subjects in the AED group who had not had significant improvement after all study assessments were completed were offered a VNS device implantation. Subjects in the VNS arm who had not had adequate improvement were evaluated for AED treatment.

Number of Subjects: Approximately 400 subjects were to be randomized at a 1:1 ratio to either AED or VNS treatment strata. Strata were to be according the AED treatment history (Early subjects were previously treated and failed treatment with 2 to 5 AEDs, Non-early subjects were treated and failed treatment with >5 AEDs). At least 15 study sites were to enroll subjects. Initially, only United Kingdom (UK) sites were to be selected. During the course of the trial, an extension was used to add non-UK centers.

A total of 151 subjects underwent screening prior to enrollment. Eight failed screening, and 143 went on to be randomized. Of those randomized, 8 subjects (4 in each of the treatment groups) were not treated. One patient in the VNS arm was explanted prior to initiation of device stimulation, so they were excluded. Therefore, 134 subjects were treated (ITT population): 65 were implanted with the VNS system and 69 were treated with AED. Nineteen investigational sites in the UK, Austria, Belgium, Germany, and Sweden participated in this study and enrolled subjects.

Study Duration: The maximum study follow-up was approximately 14 months from enrollment to study exit. The study was terminated due to insufficient enrollment prior to reaching the 400 subjects as specified in the protocol. After 4.5 years of enrollment, the Sponsor terminated enrollment and followed the remaining subjects out to the 52 week follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

1. Refractory seizures
2. Having tried at least two appropriate anti-epileptic drugs (AEDs) tested to tolerance or to blood levels at upper end of the target range of which at least 2 have been tolerated at normal dose;
3. Having at least 3 appropriate AEDs left to try
4. Having his/her current AED medication at an optimal dose at baseline
5. At least three seizures per month (average over 2 months prior to admission), excluding absences.
6. No more than four (4) weeks between seizures (over 2 months prior to admission)
7. Age 17 years or less
8. Having been evaluated for epilepsy surgery and resective surgery not felt indicated or patient/parents/legal guardian declined.
9. Patient is a male or patient is a nonpregnant female adequately protected from conception. Females of childbearing potential must use an acceptable method of birth control. Abstinence is an acceptable means of birth control
10. Patient or legal guardian understands study procedures and has voluntarily signed an informed consent in accordance with institutional policies.

Exclusion Criteria:

1. Having tried less then 2 AEDs tested to tolerance or to blood levels at upper end of the target range of which at least 2 have been tolerated at normal doses in the patient's lifetime
2. A progressive neurological condition (e.g. brain tumor etc.)
3. Inability of the parents or reluctance of the child to comply with the frequency of clinic visits during the treatment phase
4. Patient has a history of noncompliance for seizure diary completion.
5. Patient has taken an investigational drug within a period of five times the mean elimination half-life of the investigational drug plus two weeks.
6. Patient is currently using another investigational device or drug.
7. Patient is likely to require a whole body Magnetic resonance imaging (MRI) after VNS Therapy device implantation. (Refer to the Physician's Manual for the NCP Generator for additional information on the use of MRI.)
8. Patient is currently receiving or likely to receive short-wave diathermy, microwave diathermy, or therapeutic ultrasound diathermy after implantation (Refer to Physician's Manual for the VNS (Vagus Nerve Stimulation) Therapy device for additional information on the contraindicated use of diathermy).
9. Patient was previously enrolled in this or any other VNS Therapy device Study.
10. Patient has an active peptic ulcer
11. Patient has another unstable medical condition likely to precipitate seizures and make it difficult to evaluate to evaluate efficacy (e.g. diabetes)
12. Patient has had a unilateral or bilateral cervical vagotomy.
13. Patient is pregnant at the time of enrolment.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 134 (Actual)
Dates: Start 2004-10; Primary Completion 2009-12 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Bunker, PharmD, Study Director — Cyberonics, Inc.
Locations (19):
- Medical University of Vienna - Vienna General Hospital (AKH), Vienna, Austria
- ULB- Hospital Erasme, Brussels, Belgium
- Germany (2):
  - Kinderklinik der Justus-Liebig Universität, Giessen
  - University Children's Hospital, Lübeck
- Sweden (3):
  - University Hospital Lund, Lund
  - Astrid Lindgrens Barnsjukhus Karolinska, Stockholm
  - Uppsala University Hospital, Uppsala
- United Kingdom (12):
  - Birmingham Children's Hospital, Birmingham
  - Royal Hospital for Sick Children, Bristol
  - Addenbrookes Hospital, Cambridge
  - Ninewells Hospital & Medical School, Dundee
  - Leeds General Infirmary, Leeds
  - Great Ormond Street Hospital for Children, London
  - King's College Hospital, London
  - Royal Manchester Children's Hospital, Manchester
  - Sir James Spence Institute - Royal Victoria Infirmary, Newcastle
  - Queens's Medical Centre Nottingham, Nottingham
  - Sheffield Children's Hospital, Sheffield
  - Southampton Hospital, Southampton

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects selected for participation in this clinical investigation were chosen from the investigator's general subject population or were referred by a physician who knew the subject well. They were selected for inclusion after consideration of the indications and contraindications of the device. Subjects were outpatients or inpatients.
Pre-assignment Details: Subjects were randomized to VNS or AED treatment groups at a 1:1 ratio after being stratified according to their number of previous AED treatments. Of 143 randomized 8 subjects were not treated. One subject (VNS arm) was explanted before device stimulation & excluded. Therefore, 134 [actual] subjects were treated (ITT group): 65 (VNS), 69 (AED).
Groups:
- Vagus Nerve Stimulation (VNS) - ITT Population: Vagus Nerve Stimulation (VNS) Therapy
- Anti-Epileptic Drug (AED) - ITT Population: Anti-epileptic drug therapy
Period: Baseline [Visits 1 & 2]
Arm/Group | Vagus Nerve Stimulation (VNS) - ITT Population | Anti-Epileptic Drug (AED) - ITT Population
Started | 66 | 69
Actual Patients Treated | 65 | 69
Completed | 65 | 69
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0
Period: Treatment Phase (VNS/AED) [Visits 3-10]
Arm/Group | Vagus Nerve Stimulation (VNS) - ITT Population | Anti-Epileptic Drug (AED) - ITT Population
Started | 65 | 69
Completed | 65 | 69
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Vagus Nerve Stimulation (VNS) Therapy - ITT Population: Vagus Nerve Stimulation (VNS) Therapy is delivered by an implantable device similar to a pacemaker that sends mild stimulation to the left vagus nerve to help improve seizure control.
  The intent-to-treat (ITT) population, defined as all subjects in VNS Therapy arm implanted with the VNS Therapy System (and the device had been turned on), and the Non-VNS arm, defined as all subjects who took at least 1 dose of study AED.
- Anti-Epileptic Drug (AED) - ITT Population: This arm will supply a comparison between VNS and new AEDs which is necessary to determine an overall treatment regimen for the 30% to 40% of patients who fail to respond to 2 AEDs.
  The intent-to-treat (ITT) population, defined as all subjects in VNS Therapy arm implanted with the VNS Therapy System (and the device had been turned on), and the Non-VNS arm, defined as all subjects who took at least 1 dose of study AED.
- Total: Total of all reporting groups
Arm/Group | Vagus Nerve Stimulation (VNS) Therapy - ITT Population | Anti-Epileptic Drug (AED) - ITT Population | Total
Number analyzed (Participants) | 65 | 69 | 134
Age, Continuous [Mean (Standard Deviation); unit: years] — Age at Enrollment (Years)
  years | 10.7 (3.5) | 10.8 (3.4) | 10.7 (3.4)
Sex: Female, Male [Count of Participants; unit: Participants] — Treatment Group; VNS (n=65), AED (n=69), Total (n=134)
  Participants
    Female | 32 | 26 | 58
    Male | 33 | 43 | 76
Number of Failed Medications [Median (Full Range); unit: Number of failed medications] | 6.0 (2.2) [3 to 11] | 6.0 (2.4) [2 to 11] | 6.0 (2.3) [2 to 11]
Age at Epilepsy Onset (years) [Mean (Standard Deviation); unit: years] | 2.4 (2.7) | 2.7 (2.9) | 2.6 (2.8)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Responders After 1 Year of Follow-up (ITT-population)
Description: Responders are subjects who had no new AEDs added or significant dose changes in baseline AEDs within 1 year of follow-up, along with a reduction in the percentage change in seizure frequency from baseline to the 2-month period prior to the 1-year follow-up of at least 50%.
Time Frame: 52 weeks post baseline
Population: Subjects were stratified based on AED therapy history (Early: treated with 2 to 5 AEDs versus Non-early: treated with >5 AEDs).
Measure: Number; unit: percentage of responders
Groups:
- Vagus Nerve Stimulation (VNS) - Early Group: Patients who were treated with 2-5 AEDs prior to study entry who were randomized to VNS Therapy.
- Vagus Nerve Stimulation (VNS) - Non-Early Group: Patients who were treated with >5 AEDs prior to study entry who were randomized to VNS Therapy.
- Anti-Epileptic Drug (AED) - Early Group: Patients who were treated with 2-5 AEDs prior to study entry who were randomized to AED Group.
- Anti-Epileptic Drug (AED) - Non-Early Group: Patients who were treated with >5 AEDs prior to study entry who were randomized to AED Group.
Arm/Group | Vagus Nerve Stimulation (VNS) - Early Group | Vagus Nerve Stimulation (VNS) - Non-Early Group | Anti-Epileptic Drug (AED) - Early Group | Anti-Epileptic Drug (AED) - Non-Early Group
Number analyzed (Participants) | 23 | 33 | 23 | 25
percentage of responders | 21.7 (129.1) | 39.4 | 30.4 (90.9) | 24.0
Statistical Analysis 1: Comparison: Vagus Nerve Stimulation (VNS) - Early Group vs Anti-Epileptic Drug (AED) - Early Group; Test type: Superiority or Other; p = 0.507, Cochran-Mantel-Haenszel
Statistical Analysis 2: Comparison: Vagus Nerve Stimulation (VNS) - Non-Early Group vs Anti-Epileptic Drug (AED) - Non-Early Group; Test type: Superiority or Other; p = 0.220, Cochran-Mantel-Haenszel
Statistical Analysis 3: Comparison: Vagus Nerve Stimulation (VNS) - Early Group vs Vagus Nerve Stimulation (VNS) - Non-Early Group; Test type: Superiority or Other; p = 0.168, Cochran-Mantel-Haenszel
Statistical Analysis 4: Comparison: Anti-Epileptic Drug (AED) - Early Group vs Anti-Epileptic Drug (AED) - Non-Early Group; Test type: Superiority or Other; p = 0.620, Cochran-Mantel-Haenszel

2. Secondary Outcome: Mean Percent Change in Hague Seizure Severity Scale Score (ITT Population)
Description: The Hague Seizure Severity Assessment (Carpay et al. 1996) is a scale completed by the patient and/or caregiver to assess the severity and post-ictal recovery of seizures. A reduction in the HSSA score reflects less seizure severity experienced.
Time Frame: 52 weeks post baseline
Measure: Mean (Standard Deviation); unit: Percent Change
Groups:
- Vagus Nerve Stimulation (VNS) Early: Patients who were treated with 2-5 AEDs prior to study entry who were randomized to VNS Therapy.
- Vagus Nerve Stimulation (VNS) Non-Early: Patients who were treated with >5 AEDs prior to study entry who were randomized to VNS Therapy.
- Anti-Epileptic Drug (AED) Early: Patients who were treated with 2-5 AEDs prior to study entry who were randomized to AED Group.
- Anti-Epileptic Drug (AED) Non-Early: Patients who were treated with >5 AEDs prior to study entry who were randomized to AED Group.
Arm/Group | Vagus Nerve Stimulation (VNS) Early | Vagus Nerve Stimulation (VNS) Non-Early | Anti-Epileptic Drug (AED) Early | Anti-Epileptic Drug (AED) Non-Early
Number analyzed (Participants) | 25 | 32 | 24 | 27
Percent Change | -1.8 (19.1) [-30 to 50] | -7.7 (20.3) [-48 to 39] | -11.9 (17.1) [-49 to 19] | -1.4 (17.7) [-63 to 38]
Statistical Analysis 1: Comparison: Vagus Nerve Stimulation (VNS) Early vs Anti-Epileptic Drug (AED) Early; Test type: Superiority or Other; p = 0.727, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Vagus Nerve Stimulation (VNS) Non-Early vs Anti-Epileptic Drug (AED) Non-Early; Test type: Superiority or Other; p = 0.217, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Vagus Nerve Stimulation (VNS) Early vs Vagus Nerve Stimulation (VNS) Non-Early; Test type: Superiority or Other; p = 0.270, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Anti-Epileptic Drug (AED) Early vs Anti-Epileptic Drug (AED) Non-Early; Test type: Superiority or Other; p = 0.036, Wilcoxon (Mann-Whitney)

3. Secondary Outcome: Wellcome Quality of Life Assessment (Questionnaire A) in Epilepsy (ITT Population)
Description: Calculate changes in the Wellcome Quality of Life Assessment (Parker et al. 1999) (Questionnaire A) for patients in both treatment arms (AED and VNS) at 52 weeks after randomization compared to baseline. The higher the quality of life score the better the quality of life experienced.
  An analysis of variance (ANOVA) model will be used to adjust for baseline variables (including QoL score) when comparing the two treatment groups. A two-sample t-test will be used for simple comparison QoL change from baseline.
  Total range for this scale is a minimum score of 81 to a maximum score of 336. There are no applicable subscales.
Time Frame: 52 weeks post baseline
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Vagus Nerve Stimulation (VNS) - Early Group | Vagus Nerve Stimulation (VNS) - Non-Early Group | Anti-Epileptic Drug (AED) - Early Group | Anti-Epileptic Drug (AED) - Non-Early Group
Number analyzed (Participants) | 12 | 17 | 9 | 17
Scores on a Scale | 26.7 (27.1) | 30.6 (48.5) | 17.0 (29.9) | -2.1 (30.9)
Statistical Analysis 1: Comparison: Vagus Nerve Stimulation (VNS) - Early Group vs Anti-Epileptic Drug (AED) - Early Group; Test type: Superiority or Other; p = 0.448, t-test, 2 sided
Statistical Analysis 2: Comparison: Vagus Nerve Stimulation (VNS) - Non-Early Group vs Anti-Epileptic Drug (AED) - Non-Early Group; Test type: Superiority or Other; p = 0.025, t-test, 2 sided
Statistical Analysis 3: Comparison: Vagus Nerve Stimulation (VNS) - Early Group vs Vagus Nerve Stimulation (VNS) - Non-Early Group; Test type: Superiority or Other; p = 0.799, t-test, 2 sided
Statistical Analysis 4: Comparison: Anti-Epileptic Drug (AED) - Early Group vs Anti-Epileptic Drug (AED) - Non-Early Group; Test type: Superiority or Other; p = 0.142, t-test, 2 sided

4. Secondary Outcome: Hague Restriction in Childhood Epilepsy Scale (Questionnaire B) (ITT Population)
Description: Calculate changes in the Hague Restriction in Childhood Epilepsy scale (Carpay et al. 1997) (Questionnaire B) for patients in both treatment arms (AED and VNS) at 52 weeks after randomization compared to baseline. The higher the quality of life score the better the quality of life experienced.
  An analysis of variance (ANOVA) model will be used to adjust for baseline variables (including QoL score) when comparing the two treatment groups. A two-sample t-test will be used for simple comparison QoL change from baseline.
  Total range for this scale is a minimum score of 10 to a maximum score of 40. There are no applicable subscales.
Time Frame: 52 weeks post baseline
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Vagus Nerve Stimulation (VNS) - Early Group | Vagus Nerve Stimulation (VNS) - Non-Early Group | Anti-Epileptic Drug (AED) - Early Group | Anti-Epileptic Drug (AED) - Non-Early Group
Number analyzed (Participants) | 14 | 18 | 17 | 12
Scores on a Scale | 1.6 (5.6) | 3.0 (5.3) | 2.5 (7.6) | 1.3 (6.5)
Statistical Analysis 1: Comparison: Vagus Nerve Stimulation (VNS) - Early Group vs Anti-Epileptic Drug (AED) - Early Group; Test type: Superiority or Other; p = 0.714, t-test, 2 sided
Statistical Analysis 2: Comparison: Vagus Nerve Stimulation (VNS) - Non-Early Group vs Anti-Epileptic Drug (AED) - Non-Early Group; Test type: Superiority or Other; p = 0.426, t-test, 2 sided
Statistical Analysis 3: Comparison: Vagus Nerve Stimulation (VNS) - Early Group vs Vagus Nerve Stimulation (VNS) - Non-Early Group; Test type: Superiority or Other; p = 0.467, t-test, 2 sided
Statistical Analysis 4: Comparison: Anti-Epileptic Drug (AED) - Early Group vs Anti-Epileptic Drug (AED) - Non-Early Group; Test type: Superiority or Other; p = 0.654, t-test, 2 sided

5. Secondary Outcome: Mean Percent Change in Seizure Frequency (ITT Population)
Description: The mean percent change in seizure frequency for the VNS and AED treatment groups at 52 weeks post baseline.
  Both AED and VNS treatment groups were stratified according to the patients' number of previous AED treatments ("early group" had 2 to 5 AEDs tested to tolerance or to blood levels at upper end of target range; "non-early group" had more than 5 AEDs tested to tolerance or to blood levels at upper end of target range). Seizure frequency was calculated based on number of patient/caregiver reported seizures at 52-week post baseline (percentage change in seizure frequency from baseline to the 2-month period prior to the 1-year follow-up of at least 50%). All seizures were counted.
  The safety population consists of 66 VNS implanted patients and the AED safety population includes 69 patients who are randomized to the AED arm.
  Please note one patient in the VNS safety population who was implanted but never received stimulation was excluded from the ITT population.
Time Frame: 52 weeks post baseline
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Vagus Nerve Stimulation (VNS) Early | Vagus Nerve Stimulation (VNS) Non-Early | Anti-Epileptic Drug (AED) Early | Anti-Epileptic Drug (AED) Non-Early
Number analyzed (Participants) | 23 | 33 | 23 | 25
Percent Change | 28.6 (177.5) | -5.0 (80.7) | 10.5 (123.2) | -17.3 (43.3)
Statistical Analysis 1: Comparison: Vagus Nerve Stimulation (VNS) Early vs Anti-Epileptic Drug (AED) Early; Test type: Superiority or Other; p = 0.691, ANOVA
Statistical Analysis 2: Comparison: Vagus Nerve Stimulation (VNS) Non-Early vs Anti-Epileptic Drug (AED) Non-Early; Test type: Superiority or Other; p = 0.494, ANOVA
Statistical Analysis 3: Comparison: Vagus Nerve Stimulation (VNS) Early vs Vagus Nerve Stimulation (VNS) Non-Early; Test type: Superiority or Other; p = 0.343, ANOVA
Statistical Analysis 4: Comparison: Anti-Epileptic Drug (AED) Early vs Anti-Epileptic Drug (AED) Non-Early; Test type: Superiority or Other; p = 0.295, ANOVA

6. Secondary Outcome: Number of Subjects With Any Non-Serious Adverse Events by System Organ Class and Preferred Term (Safety Population)
Description: To compare the safety of Vagus Nerve Stimulation (VNS) treatment using the VNS Therapy device to anti-epileptic drug (AED) therapy in treating patients with seizures.
  The safety population consists of 66 VNS implanted patients and the AED safety population includes 69 patients who are randomized to the AED arm.
  Please note one patient in the VNS safety population who was implanted but never received stimulation was excluded from the ITT population.
Time Frame: 0-52 weeks
Population: Number of participants with any definite related Adverse Event by body system and preferred term, Safety Population.
  NOTE: Number of participants analyzed in VNS arm includes one explant not from ITT population, but from safety population.
Measure: Number; unit: Participants
Groups:
- Vagus Nerve Stimulation (VNS): Patients who were either treated with >5 AEDs or treated with 2-5 AEDs prior to study entry and were randomized to VNS Therapy.
- Anti-Epileptic Drug (AED): Patients who were either treated with >5 AEDs or treated with 2-5 AEDs prior to study entry and were randomized to AED Group.
Arm/Group | Vagus Nerve Stimulation (VNS) | Anti-Epileptic Drug (AED)
Number analyzed (Participants) | 66 | 69
Participants
  Blood and lymphatic system disorders | 0 | 1
  Eye disorders | 0 | 1
  Gastrointestinal disorders | 1 | 4
  Ear and labyrinth disorders | 1 | 0
  Infections and infestations | 4 | 0
  Nervous system disorders | 6 | 6
  Psychiatric disorders | 1 | 6
  Respiratory and mediastinal disorders | 5 | 2
  Skin and subcutaneous tissue disorders | 1 | 2
  General disorders & administration site conditions | 2 | 0
  Injury, poisoning and procedural complications | 0 | 2
  Investigations - weight decreased | 0 | 1
  Metabolism and nutrition disorders | 2 | 2
  Musculoskeletal & connective tissue disorders | 1 | 1

7. Secondary Outcome: Number of Subjects With Any Serious Adverse Events by System Organ Class & Preferred Term (Safety Population)
Description: as for outcome 6
Time Frame: 0-52 weeks
Measure: Number; unit: participants
Arm/Group | Vagus Nerve Stimulation (VNS) | Anti-Epileptic Drug (AED)
Number analyzed (Participants) | 66 | 69
participants
  Infections and infestations | 1 | 2
  Injury, poisoning and procedural complications | 0 | 2
  Nervous system disorders | 2 | 7
  Skin and subcutaneous tissue disorders | 1 | 1
  Surgical and medical procedures | 2 | 5

ADVERSE EVENTS:
Time Frame: 0-52 Weeks (1-Year)
Description: The safety population consists of 66 VNS implanted patients and the AED safety population includes 69 patients who are randomized to the AED arm.
  Please note one patient in the VNS safety population who was implanted but never received stimulation was excluded from the ITT population.
Groups:
- Vagus Nerve Stimulation (VNS) Therapy - Safety Population: Vagus Nerve Stimulation (VNS) Therapy is delivered by an implantable device similar to a pacemaker that sends mild stimulation to the left vagus nerve to help improve seizure control.
  All subjects were considered evaluable for tolerability and safety after implantation of the VNS Therapy System.
  NOTE: Number of participants analyzed in VNS safety population includes one patient explanted that did not receive stimulation and was therefore excluded from ITT population.
- Anti-Epileptic Drug (AED) - Safety Population: This arm will supply a comparison between VNS and new AEDs which is necessary to determine an overall treatment regimen for the 30% to 40% of patients who fail to respond to 2 AEDs.
  All subjects were considered evaluable for tolerability and safety after initiation of adjunctive AED treatment.
Arm/Group | Vagus Nerve Stimulation (VNS) Therapy - Safety Population | Anti-Epileptic Drug (AED) - Safety Population
Serious Adverse Events (participants affected / at risk) | 5/66 | 10/69
Other Adverse Events (participants affected / at risk) | 20/66 | 25/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vagus Nerve Stimulation (VNS) Therapy - Safety Population (N=66) | Anti-Epileptic Drug (AED) - Safety Population (N=69)
Tonsilitis (Infections and infestations) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 2 (2) | 5 (5)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Adenoidectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Status epilepticus (Nervous system disorders) | 0 (0) | 2 (2)
Stevens Johnson Syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hospitalization (Surgical and medical procedures) | 0 (0) | 3 (3)
Investigation (Surgical and medical procedures) | 0 (0) | 1 (1)
Medical device removal (Surgical and medical procedures) | 1 (1) | 0 (0)
Surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Tonsillectomy (Surgical and medical procedures) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vagus Nerve Stimulation (VNS) Therapy - Safety Population (N=66) | Anti-Epileptic Drug (AED) - Safety Population (N=69)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
External ear disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1)
Abdonimal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2)
Fatigue (General disorders) | 1 (1) | 0 (0)
Localised oedema (General disorders) | 1 (1) | 0 (0)
Medical device pain (General disorders) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 2 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Convulsion (Nervous system disorders) | 2 (2) | 4 (4)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Dysarthia (Nervous system disorders) | 0 (0) | 1 (1)
Grand mal convulsion (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
Myoclonus (Nervous system disorders) | 1 (1) | 0 (0)
Psychomotor hyperactivity (Nervous system disorders) | 2 (2) | 0 (0)
Sedation (Nervous system disorders) | 0 (0) | 2 (2)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Speech disorder (Nervous system disorders) | 1 (1) | 0 (0)
Abnormal behavior (Psychiatric disorders) | 0 (0) | 3 (3)
Breath holding (Psychiatric disorders) | 0 (0) | 1 (1)
Depressed mood (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin nodule (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Study was terminated due to low enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days